CLINICAL TRIAL: NCT03292185
Title: A Single Centre, Randomised, Double-blind, Three-period Cross-over Trial to Investigate the Single Dose Pharmacokinetics of Insulin Degludec/Liraglutide Compared With Insulin Degludec and Liraglutide in Healthy Chinese Subjects
Brief Title: A Trial to Investigate the Single Dose Pharmacokinetics of Insulin Degludec/Liraglutide Compared With Insulin Degludec and Liraglutide in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9068-4139; U1111-1155-0990 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec; Liraglutide

STUDY DESIGN:
Intervention Model Description: Three-period complete cross-over, six treatment sequences
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- IDeglira-IDeg-Liraglutide (Experimental): Treatment sequence first Insulin Degludec/Liraglutide, then Insulin Degludec, then Liraglutide
  Interventions: Drug: insulin degludec/liraglutide; Drug: insulin degludec; Drug: liraglutide
- IDeglira-Liraglutide-IDeg (Experimental): Treatment sequence first Insulin Degludec/Liraglutide, then Liraglutide, then Insulin Degludec
  Interventions: Drug: insulin degludec/liraglutide; Drug: insulin degludec; Drug: liraglutide
- IDeg-Liraglutide-IDeglira (Experimental): Treatment sequence first Isulin Degludec, then Liraglutide, then Insulin Degludec/Liraglutide
  Interventions: Drug: insulin degludec/liraglutide; Drug: insulin degludec; Drug: liraglutide
- IDeg-IDeglira-Liraglutide (Experimental): Treatment sequence first Insulin Degludec, then Insulin Degludec/Liraglutide, then Liraglutide
  Interventions: Drug: insulin degludec/liraglutide; Drug: insulin degludec; Drug: liraglutide
- Liraglutide-IDeg-IDeglira (Experimental): Treatment sequence first Liraglutide, then Insulin Degludec, then Insulin Degludec/Liraglutide
  Interventions: Drug: insulin degludec/liraglutide; Drug: insulin degludec; Drug: liraglutide
- Liraglutide-IDeglira-IDeg (Experimental): Treatment sequence first Liraglutide, then Insulin Degludec/Liraglutide, then Insulin Degludec
  Interventions: Drug: insulin degludec/liraglutide; Drug: insulin degludec; Drug: liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Insulin Degludec/Liraglutide combination product with 0.61 mg Liraglutide and 17 U Insulin Degludec, single dose administration under the skin in the thigh.
Drug: insulin degludec — 17 U Insulin Degludec, single dose administration under the skin in the thigh.
Drug: liraglutide — 0.6 mg Liraglutide, single dose administration under the skin in the thigh

SUMMARY:
The main purpose of the trial is to compare the bioavailability (extent of drug absorption into the circulation) of insulin degludec and liraglutide as part of a combination product insulin degludec/liraglutide compared to the corresponding doses of single, separate injections of insulin degludec and liraglutide. Participants will receive all three test substances. The order of trial administration will be allocated by chance. During the trial period, serials of blood samples will be collected from the participants at three dosing periods, in order to determine the concentration of insulin degludec and liraglutide. The total volume of blood taken throughout the whole trial period will be less than 400 mL. Participants will be asked to stay on daytime and overnight in the trial sites on some predefined days. For other outpatient days, participants need to attend the trial site as required for drug administration or required assessments.

ELIGIBILITY:
Inclusion criteria:

* Male and female Chinese subjects, who are considered to be generally healthy, based on assessment of medical history, physical examination, and clinical laboratory data, as judged by the investigator
* Age between 18 to 45 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 19.0 and 24.0 kg/sqm (both inclusive)
* Body weight at least 50.0 kg
* Fasting plasma glucose less than 6.1 mmol/L (110 mg/dL)

Exclusion criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential not using an adequate contraceptive methods throughout the trial including follow-up period. Adequate contraceptive measures are sterilisation, intrauterine device (IUD), oral contraceptives or barrier methods
* Donation of any blood or plasma in the past month or in excess of 400 mL within the 90 days preceding screening or surgery or trauma with more than 400 mL blood loss within the 90 days preceding screening
* History or presence of cancer, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrine (incl. diabetes and recurrent hypoglycaemia), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders that might have impact on the trial result, as judged by the investigator
* Use of any prescription or non-prescription medication, except for paracetamol, acetylsalicylic acid, contraceptives and vitamins (mega-dose vitamin therapy not allowed, dose judged by the investigator) within 2 weeks prior to screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration time curve | From 0 to last quantifiable observation after single dose of insulin degludec/liraglutide and insulin degludec, assessments from 0 hours to 120 hours
  Calculated based on insulin degludec concentration in serum
Area under the plasma liraglutide concentration time curve | from 0 to last quantifiable observation after single dose of insulin degludec/liraglutide and liraglutide, assessments from 0 hours to 72 hours
  Calculated based on liraglutide concentration in plasma

SECONDARY OUTCOMES:
Area under the serum insulin degludec concentration time curve from 0 to infinity after single dose | 0 hours to 120 hours
  Calculated based on insulin degludec measured in serum
Maximum observed serum insulin degludec concentration | 0 hours to 120 hours
  Calculated based on insulin degludec measured in serum
Time to maximum serum insulin degludec concentration | 0 hours to 120 hours
  Calculated based on insulin degludec measured in serum
Terminal elimination half-life for insulin degludec | 0 hours to 120 hours
  Calculated based on insulin degludec measured in serum
Area under the plasma liraglutide concentration time curve from 0 to infinity after single dose | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Maximum observed plasma liraglutide concentration | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Time to maximum plasma liraglutide concentration | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Terminal elimination half-life of liraglutide | 0 hours to 72 hours
  Calculated based on liraglutide measured in plasma
Number of treatment emergent adverse events | Visit 2 (Day 1, randomisation), Visit 5 (7-14 days after last dosing visit)
  Count
Number of treatment emergent hypoglycaemic episodes | Visit 2 (Day 1, randomisation), Visit 5 (7-14 days after last dosing visit)
  Count
Local tolerability at the injection site | Visit 2 (Day 1, randomisation), Visit 5 (7-14 days after last dosing visit)
  Count

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com